CLINICAL TRIAL: NCT01667731
Title: A Phase 3, Open-label Study to Investigate the Efficacy and Safety of GS-7977 Plus Ribavirin in Chronic Genotype 1, 2 and 3 Hepatitis C Virus (HCV) and Human Immunodeficiency Virus (HIV) Co-infected Subjects
Brief Title: Efficacy and Safety of Sofosbuvir Plus Ribavirin in Chronic Genotype 1, 2 and 3 Hepatitis C Virus (HCV) and Human Immunodeficiency Virus (HIV) Co-infected Adults
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Gilead Sciences (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GS-US-334-0123
Record Dates: First submitted 2012-08-09; First posted 2012-08-17 (Estimated); Results first posted 2014-11-21 (Estimated); Last update posted 2014-11-21 (Estimated); Status verified 2014-11

CONDITIONS: Hepatitis C; Human Immunodeficiency Virus
Keywords: Hepatitis C; Chronic; HCV; HIV; Human Immunodeficiency Virus; Co-Infected
MeSH Terms: conditions — Hepatitis C; Acquired Immunodeficiency Syndrome; Bronchiolitis Obliterans Syndrome | interventions — Sofosbuvir

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- SOF+RBV 12 Weeks (GT 2/3, TN) (Experimental): Treatment-naive (TN) participants coinfected with HIV-1 and genotype (GT) 2 or genotype 3 HCV infection will receive SOF+RBV for 12 weeks.
  Interventions: Drug: SOF; Drug: RBV
- SOF+RBV 24 Weeks (GT 2/3, TE) (Experimental): Treatment-experienced (TE) participants coinfected with HIV-1 and genotype 2 or genotype 3 HCV infection will receive SOF+RBV for 24 weeks.
  Interventions: Drug: SOF; Drug: RBV
- SOF+RBV 24 Weeks (GT 1, TN) (Experimental): Treatment-naive (TN) participants coinfected with HIV-1 and genotype 1 HCV infection will receive SOF+RBV for 24 weeks.
  Interventions: Drug: SOF; Drug: RBV

INTERVENTIONS:
Drug: SOF — Sofosbuvir (SOF) 400 mg tablet administered orally once daily
  Other Names: GS-7977; PSI-7977; Sovaldi®
Drug: RBV — Ribavirin (RBV) tablets administered orally in a divided daily dose according to package insert weight-based dosing recommendations (< 75kg = 1000 mg and ≥ 75 kg = 1200 mg)

SUMMARY:
This study will evaluate the efficacy, safety, and tolerability of sofosbuvir (SOF; GS-7977) plus ribavirin (RBV) in adults with chronic genotypes 1, 2, and 3 HCV infection who are coinfected with HIV-1.

ELIGIBILITY:
Inclusion Criteria:

* Willing and able to provide written informed consent
* Male or female, age ≥ 18 years with chronic HCV and HIV-1 infection
* HCV RNA > 1 x 10^4 IU/mL at screening
* Infection with HCV genotype 1, 2 or 3 as determined at screening
* HIV-1 infection confirmed with positive ELISA or Western blot at screening
* Medical records must be sufficient to be categorized on interferon (IFN) eligibility or prior treatment history with PEG/RBV.
* Confirmation of chronic HCV infection
* Ability to determine presence/absence of cirrhosis.
* HIV antiretroviral therapy (ARV) criteria of one of the following:

  * ARV untreated with a CD4 T-cell count > 500 cells/mm^3
  * On a stable, protocol-approved, ARV for > 8 weeks prior to screening with a CD4 T-cell count > 200 cells/mm^3 and a documented undetectable plasma HIV-1 RNA level for ≥ 8 weeks preceding the screening visit
* Approved HIV antiretroviral medications based on drug interaction studies
* Not been treated with any investigational drug or device within 30 days of the screening visit
* Females if confirmed that she is not pregnant or nursing of non-childbearing potential or of childbearing potential but has a negative serum pregnancy test at screening and agrees to use protocol approved method of birth control from screening through 6 months after the last dose of RBV
* Males who agree to consistently and correctly use a condom while their female partner agrees to use protocol approved method of birth control from screening through 7 months after the last dose of RBV
* Must be of generally good health as determined by the investigator.
* Liver imaging within 6 months of baseline/Day 1 is required in cirrhotic patients only, to exclude hepatocellular carcinoma (HCC)

Exclusion Criteria:

* Non-genotype 1/2/3 or mixed genotype at screening
* Genotype 1 with prior treatment for HCV
* Poor control with ARV regimen
* Prior exposure to a direct-acting antiviral targeting the HCV nonstructural protein (NS)5B polymerase
* Chronic liver disease of a non-HCV etiology (eg, hemochromatosis, Wilson's disease, α1 antitrypsin deficiency, cholangitis)
* A new AIDS-defining condition diagnosed within 30 days prior to screening
* Active, serious infection (other than HIV or HCV) requiring parenteral antibiotics, antivirals or antifungals within 30 days prior to baseline
* Infection with hepatitis B virus (HBV)
* Contraindication to RBV therapy
* Chronic use of systemically administered immunosuppressive agents (eg, prednisone equivalent > 10 mg/day)
* History of solid organ transplantation or malignancy diagnosed or treated within 5 years
* Current or prior history of clinical hepatic decompensation or other significant gastrointestinal disorder

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 224 (Actual)
Dates: Start 2012-07; Primary Completion 2013-11 (Actual); Study Completion 2014-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Anuj Gaggar, MD, PhD, Study Director — Gilead Sciences
Locations (27):
- United States (26):
  - Birmingham, Alabama
  - Coronado, California
  - Los Angeles, California
  - Lutherville, California
  - Oakland, California
  - Sacramento, California
  - San Francisco, California
  - Torrance, California
  - Washington D.C., District of Columbia
  - Miami, Florida
  - Orlando, Florida
  - Tampa, Florida
  - Chicago, Illinois
  - Springfield, Massachusetts
  - Kansas City, Missouri
  - Hillsborough, New Jersey
  - Santa Fe, New Mexico
  - New York, New York
  - Chapel Hill, North Carolina
  - Durham, North Carolina
  - Allentown, Pennsylvania
  - Philadelphia, Pennsylvania
  - Providence, Rhode Island
  - Dallas, Texas
  - Houston, Texas
  - Seattle, Washington
- San Juan, Puerto Rico

REFERENCES:
- [Derived] Saeed S, Strumpf EC, Walmsley SL, Rollet-Kurhajec K, Pick N, Martel-Laferriere V, Hull M, Gill MJ, Cox J, Cooper C, Klein MB; Canadian Co-Infection Cohort Study; Cohen J, Conway B, Cooper C, Cote P, Cox J, Gill J, Haider S, Harris M, Haase D, Hull M, Montaner J, Moodie E, Pick N, Rachlis A, Rouleau D, Sandre R, Tyndall JM, Vachon ML, Walmsley S, Wong D. How Generalizable Are the Results From Trials of Direct Antiviral Agents to People Coinfected With HIV/HCV in the Real World? Clin Infect Dis. 2016 Apr 1;62(7):919-926. doi: 10.1093/cid/civ1222. Epub 2016 Jan 6. PMID 26743093
- [Derived] Younossi ZM, Stepanova M, Sulkowski M, Naggie S, Puoti M, Orkin C, Hunt SL. Sofosbuvir and Ribavirin for Treatment of Chronic Hepatitis C in Patients Coinfected With Hepatitis C Virus and HIV: The Impact on Patient-Reported Outcomes. J Infect Dis. 2015 Aug 1;212(3):367-77. doi: 10.1093/infdis/jiv005. Epub 2015 Jan 12. PMID 25583164
- [Derived] Sulkowski MS, Naggie S, Lalezari J, Fessel WJ, Mounzer K, Shuhart M, Luetkemeyer AF, Asmuth D, Gaggar A, Ni L, Svarovskaia E, Brainard DM, Symonds WT, Subramanian GM, McHutchison JG, Rodriguez-Torres M, Dieterich D; PHOTON-1 Investigators. Sofosbuvir and ribavirin for hepatitis C in patients with HIV coinfection. JAMA. 2014 Jul 23-30;312(4):353-61. doi: 10.1001/jama.2014.7734. PMID 25038354

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled at a total of 34 study sites in the United States. The first participant was screened on 20 July 2012. The last participant observation occurred on 10 February 2014.
Pre-assignment Details: 330 participants were screened.
Groups:
- SOF+RBV 12 Wk GT 2 TN: Sofosbuvir (SOF) 400 mg tablet once daily + ribavirin (RBV) tablets (1000-1200 mg daily based on weight) for 12 weeks (treatment naive (TN), genotype (GT) 2)
- SOF+RBV 12 Wk GT 3 TN: SOF 400 mg tablet once daily + RBV tablets (1000-1200 mg daily based on weight) for 12 weeks (treatment naive, genotype 3)
- SOF+RBV 24 Wk GT 2 TE: SOF 400 mg tablet once daily + RBV tablets (1000-1200 mg daily based on weight) for 24 weeks (treatment experienced (TE), genotype 2)
- SOF+RBV 24 Wk GT 3 TE: SOF 400 mg tablet once daily + RBV tablets (1000-1200 mg daily based on weight) for 24 weeks (treatment experienced, genotype 3)
- SOF+RBV 24 Wk GT 1 TN: SOF 400 mg tablet once daily + RBV tablets (1000-1200 mg daily based on weight) for 24 weeks (treatment naive, genotype 1)
Period: Overall Study
Arm/Group | SOF+RBV 12 Wk GT 2 TN | SOF+RBV 12 Wk GT 3 TN | SOF+RBV 24 Wk GT 2 TE | SOF+RBV 24 Wk GT 3 TE | SOF+RBV 24 Wk GT 1 TN
Started | 26 | 42 | 24 | 17 | 115
Completed | 21 | 26 | 22 | 15 | 87
Not Completed | 5 | 16 | 2 | 2 | 28
Not completed — Enrolled but not treated | 0 | 0 | 0 | 0 | 1
Not completed — Efficacy Failure | 1 | 12 | 0 | 1 | 24
Not completed — Lost to Follow-up | 2 | 3 | 1 | 1 | 2
Not completed — Subject Withdrew Consent | 2 | 0 | 1 | 0 | 1
Not completed — Death | 0 | 1 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Safety Analysis Set: participants who were enrolled and received at least 1 dose of study drug
Groups:
- SOF+RBV 12 Wk GT 2 TN: SOF 400 mg tablet once daily + RBV tablets (1000-1200 mg daily based on weight) for 12 weeks (treatment naive, genotype 2)
- SOF+RBV 24 Wk GT 2 TE: SOF 400 mg tablet once daily + RBV tablets (1000-1200 mg daily based on weight) for 24 weeks (treatment experienced, genotype 2)
- Total: Total of all reporting groups
Arm/Group | SOF+RBV 12 Wk GT 2 TN | SOF+RBV 12 Wk GT 3 TN | SOF+RBV 24 Wk GT 2 TE | SOF+RBV 24 Wk GT 3 TE | SOF+RBV 24 Wk GT 1 TN | Total
Number analyzed (Participants) | 26 | 42 | 24 | 17 | 114 | 223
Age, Continuous [Mean (Standard Deviation); unit: years] | 51 (9.7) | 48 (9.6) | 54 (4.9) | 54 (7.0) | 48 (8.4) | 49 (8.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 8 | 1 | 3 | 21 | 38
  Male | 21 | 34 | 23 | 14 | 93 | 185
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 8 | 11 | 5 | 5 | 25 | 54
  Not Hispanic or Latino | 18 | 31 | 19 | 12 | 89 | 169
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0
Race/Ethnicity, Customized [Number; unit: participants]
  Black or African American | 6 | 2 | 6 | 1 | 37 | 52
  White | 18 | 36 | 17 | 15 | 70 | 156
  Asian | 0 | 1 | 1 | 0 | 1 | 3
  American Indian/Alaska Native/First Nations | 0 | 0 | 0 | 1 | 0 | 1
  Hawaiian or Other Pacific Islander | 1 | 0 | 0 | 0 | 1 | 2
  Other | 1 | 3 | 0 | 0 | 5 | 9
HCV Genotype [Number; unit: participants]
  Genotype 1 | 0 | 0 | 0 | 0 | 114 | 114
  Genotype 2 | 26 | 0 | 24 | 0 | 0 | 50
  Genotype 3 | 0 | 42 | 0 | 17 | 0 | 59
Liver Cirrhosis [Number; unit: participants]
  No | 25 | 36 | 20 | 11 | 109 | 201
  Yes | 1 | 6 | 4 | 6 | 5 | 22
IL28b Status [Number; unit: participants] — CC, CT, and TT alleles are different forms of the IL28b gene.
  participants
    CC | 10 | 15 | 10 | 10 | 30 | 75
    CT | 15 | 22 | 10 | 7 | 57 | 111
    TT | 1 | 5 | 4 | 0 | 26 | 36
    Missing | 0 | 0 | 0 | 0 | 1 | 1
HCV RNA (log10 IU/mL) [Mean (Standard Deviation); unit: log10 IU/mL] | 6.5 (0.59) | 6.2 (0.59) | 6.5 (0.82) | 6.4 (0.47) | 6.6 (0.83) | 6.5 (0.75)
HCV RNA Category [Number; unit: participants]
  < 6 log10 IU/mL | 6 | 15 | 5 | 2 | 22 | 50
  ≥ 6 log10 IU/mL | 20 | 27 | 19 | 15 | 92 | 173

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Sustained Virologic Response (SVR) at 12 Weeks After Discontinuation of Therapy (SVR12)
Description: SVR12 was defined as HCV RNA < the lower limit of quantitation (LLOQ; ie, 25 IU/mL) at 12 weeks after stopping study treatment.
Time Frame: Posttreatment Week 12
Population: Full Analysis Set: participants who were enrolled and received at least 1 dose of study drug
Measure: Number; unit: percentage of participants
Arm/Group | SOF+RBV 12 Wk GT 2 TN | SOF+RBV 12 Wk GT 3 TN | SOF+RBV 24 Wk GT 2 TE | SOF+RBV 24 Wk GT 3 TE | SOF+RBV 24 Wk GT 1 TN
Number analyzed (Participants) | 26 | 42 | 24 | 17 | 114
percentage of participants | 88.5 | 66.7 | 91.7 | 94.1 | 76.3

2. Primary Outcome: Incidence of Adverse Events Leading to Permanent Discontinuation of Study Drug(s)
Description: The percentage of participants discontinuing any study drug due to an adverse event was summarized.
Time Frame: Up to 24 weeks
Population: Safety Analysis Set: participants who were enrolled and received at least 1 dose of study drug
Measure: Number; unit: percentage of participants
Groups:
- SOF+RBV 12 Wk GT 2/3 TN: SOF 400 mg tablet once daily + RBV tablets (1000-1200 mg daily based on weight) for 12 weeks (treatment naive, genotypes 2 and 3)
- SOF+RBV 24 Wk GT 2/3 TE: SOF 400 mg tablet once daily + RBV tablets (1000-1200 mg daily based on weight) for 24 weeks (treatment experienced, genotypes 2 and 3)
Arm/Group | SOF+RBV 12 Wk GT 2/3 TN | SOF+RBV 24 Wk GT 2/3 TE | SOF+RBV 24 Wk GT 1 TN
Number analyzed (Participants) | 68 | 41 | 114
percentage of participants | 4.4 | 2.4 | 2.6

3. Secondary Outcome: Percentage of Participants With Sustained Virologic Response at 4 and 24 Weeks After Discontinuation of Therapy (SVR4 and SVR24)
Description: SVR4 and SVR24 were defined as HCV RNA < LLOQ at 4 and 24 weeks following the last dose of study drug, respectively.
Time Frame: Posttreatment Weeks 4 and 24
Population: Full Analysis Set
Measure: Number; unit: percentage of participants
Arm/Group | SOF+RBV 12 Wk GT 2 TN | SOF+RBV 12 Wk GT 3 TN | SOF+RBV 24 Wk GT 2 TE | SOF+RBV 24 Wk GT 3 TE | SOF+RBV 24 Wk GT 1 TN
Number analyzed (Participants) | 26 | 42 | 24 | 17 | 114
percentage of participants
  SVR4 | 88.5 | 71.4 | 95.8 | 94.1 | 80.7
  SVR24 | 88.5 | 66.7 | 91.7 | 88.2 | 75.4

4. Secondary Outcome: Change From Baseline in HCV RNA at Week 1
Time Frame: Baseline; Week 1
Population: Participants in the Full Analysis Set with available data were analyzed.
Measure: Mean (Standard Deviation); unit: log10 IU/mL
Arm/Group | SOF+RBV 12 Wk GT 2 TN | SOF+RBV 12 Wk GT 3 TN | SOF+RBV 24 Wk GT 2 TE | SOF+RBV 24 Wk GT 3 TE | SOF+RBV 24 Wk GT 1 TN
Number analyzed (Participants) | 25 | 40 | 24 | 16 | 108
log10 IU/mL | -4.69 (0.471) | -4.52 (0.464) | -4.63 (0.680) | -4.78 (0.354) | -4.42 (0.958)

5. Secondary Outcome: Change From Baseline in HCV RNA at Week 2
Time Frame: Baseline; Week 2
Population: Participants in the Full Analysis Set with available data were analyzed.
Measure: Mean (Standard Deviation); unit: log10 IU/mL
Arm/Group | SOF+RBV 12 Wk GT 2 TN | SOF+RBV 12 Wk GT 3 TN | SOF+RBV 24 Wk GT 2 TE | SOF+RBV 24 Wk GT 3 TE | SOF+RBV 24 Wk GT 1 TN
Number analyzed (Participants) | 26 | 41 | 24 | 17 | 112
log10 IU/mL | -5.11 (0.574) | -4.84 (0.579) | -5.15 (0.813) | -5.06 (0.467) | -5.00 (0.829)

6. Secondary Outcome: Change From Baseline in HCV RNA at Week 4
Time Frame: Baseline; Week 4
Population: Participants in the Full Analysis Set with available data were analyzed.
Measure: Mean (Standard Deviation); unit: log10 IU/mL
Arm/Group | SOF+RBV 12 Wk GT 2 TN | SOF+RBV 12 Wk GT 3 TN | SOF+RBV 24 Wk GT 2 TE | SOF+RBV 24 Wk GT 3 TE | SOF+RBV 24 Wk GT 1 TN
Number analyzed (Participants) | 26 | 41 | 24 | 17 | 114
log10 IU/mL | -5.04 (0.710) | -4.86 (0.602) | -5.16 (0.820) | -5.06 (0.467) | -5.12 (0.957)

7. Secondary Outcome: Change From Baseline in HCV RNA at Week 6
Time Frame: Baseline; Week 6
Population: Participants in the Full Analysis Set with available data were analyzed.
Measure: Mean (Standard Deviation); unit: log10 IU/mL
Arm/Group | SOF+RBV 12 Wk GT 2 TN | SOF+RBV 12 Wk GT 3 TN | SOF+RBV 24 Wk GT 2 TE | SOF+RBV 24 Wk GT 3 TE | SOF+RBV 24 Wk GT 1 TN
Number analyzed (Participants) | 26 | 41 | 24 | 17 | 110
log10 IU/mL | -5.13 (0.593) | -4.86 (0.602) | -5.16 (0.820) | -5.06 (0.467) | -5.20 (0.785)

8. Secondary Outcome: Change From Baseline in HCV RNA at Week 8
Time Frame: Baseline; Week 8
Population: Participants in the Full Analysis Set with available data were analyzed.
Measure: Mean (Standard Deviation); unit: log10 IU/mL
Arm/Group | SOF+RBV 12 Wk GT 2 TN | SOF+RBV 12 Wk GT 3 TN | SOF+RBV 24 Wk GT 2 TE | SOF+RBV 24 Wk GT 3 TE | SOF+RBV 24 Wk GT 1 TN
Number analyzed (Participants) | 26 | 40 | 24 | 17 | 111
log10 IU/mL | -5.13 (0.593) | -4.83 (0.589) | -5.16 (0.820) | -5.06 (0.467) | -5.20 (0.785)

9. Secondary Outcome: Percentage of Participants Experiencing On-treatment Virologic Failure
Description: On-treatment virologic failure was defined as:
  1. Viral breakthrough: HCV RNA ≥ LLOQ after having previously had HCV RNA < LLOQ while on treatment, confirmed with 2 consecutive values (second confirmation value may have been posttreatment) or with a last available on-treatment measurement and no subsequent follow-up values, or
  2. Viral rebound: > 1 log10 IU/mL increase in HCV RNA from nadir while on treatment, confirmed with 2 consecutive values (second confirmation value may have been posttreatment) or with a last available on-treatment measurement and no subsequent follow-up values, or
  3. Nonresponse: HCV RNA persistently ≥ LLOQ through 8 weeks of treatment
Time Frame: Up to 24 weeks
Population: Full Analysis Set
Measure: Number; unit: percentage of participants
Arm/Group | SOF+RBV 12 Wk GT 2 TN | SOF+RBV 12 Wk GT 3 TN | SOF+RBV 24 Wk GT 2 TE | SOF+RBV 24 Wk GT 3 TE | SOF+RBV 24 Wk GT 1 TN
Number analyzed (Participants) | 26 | 42 | 24 | 17 | 114
percentage of participants | 3.8 | 0 | 0 | 0 | 0.9

10. Secondary Outcome: Percentage of Participants Experiencing Viral Relapse
Description: Viral relapse was defined as having achieved undetectable HCV RNA levels (HCV RNA < LLOQ) at end of treatment, but did not achieve an SVR.
Time Frame: Up to Posttreatment Week 24
Population: Participants in the Full Analysis Set with available data were analyzed.
Measure: Number; unit: percentage of participants
Arm/Group | SOF+RBV 12 Wk GT 2 TN | SOF+RBV 12 Wk GT 3 TN | SOF+RBV 24 Wk GT 2 TE | SOF+RBV 24 Wk GT 3 TE | SOF+RBV 24 Wk GT 1 TN
Number analyzed (Participants) | 25 | 42 | 24 | 17 | 113
percentage of participants | 0 | 28.6 | 4.2 | 5.9 | 22.1

ADVERSE EVENTS:
Time Frame: Up to 24 weeks plus 30 days
Description: Safety Analysis Set
Arm/Group | SOF+RBV 12 Wk GT 2/3 TN | SOF+RBV 24 Wk GT 2/3 TE | SOF+RBV 24 Wk GT 1 TN
Serious Adverse Events (participants affected / at risk) | 5/68 | 1/41 | 8/114
Other Adverse Events (participants affected / at risk) | 57/68 | 37/41 | 106/114
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | SOF+RBV 12 Wk GT 2/3 TN (N=68) | SOF+RBV 24 Wk GT 2/3 TE (N=41) | SOF+RBV 24 Wk GT 1 TN (N=114)
Anaemia (Blood and lymphatic system disorders) | 0 | 0 | 1
Leukocytosis (Blood and lymphatic system disorders) | 0 | 0 | 1
Atrial fibrillation (Cardiac disorders) | 0 | 0 | 1
Atrial flutter (Cardiac disorders) | 0 | 0 | 1
Acute myocardial infarction (Cardiac disorders) | 1 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 1
Colitis (Gastrointestinal disorders) | 0 | 0 | 1
Enteritis (Gastrointestinal disorders) | 0 | 0 | 1
Chest pain (General disorders) | 0 | 0 | 1
Cellulitis (Infections and infestations) | 0 | 0 | 2
Pneumonia (Infections and infestations) | 1 | 1 | 0
Gastroenteritis salmonella (Infections and infestations) | 0 | 0 | 1
Respiratory tract infection (Infections and infestations) | 0 | 0 | 1
Incision site infection (Infections and infestations) | 1 | 0 | 0
Septic shock (Infections and infestations) | 1 | 0 | 0
Staphylococcal bacteraemia (Infections and infestations) | 1 | 0 | 0
Intentional overdose (Injury, poisoning and procedural complications) | 1 | 0 | 1
Fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 0 | 0 | 1
Altered state of consciousness (Nervous system disorders) | 0 | 0 | 1
Encephalopathy (Nervous system disorders) | 1 | 0 | 0
Bipolar disorder (Psychiatric disorders) | 0 | 0 | 1
Completed suicide (Psychiatric disorders) | 1 | 0 | 0
Drug abuse (Psychiatric disorders) | 1 | 0 | 0
Suicide attempt (Psychiatric disorders) | 1 | 0 | 0
Renal failure acute (Renal and urinary disorders) | 1 | 0 | 2
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Leukocytoclastic vasculitis (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | SOF+RBV 12 Wk GT 2/3 TN (N=68) | SOF+RBV 24 Wk GT 2/3 TE (N=41) | SOF+RBV 24 Wk GT 1 TN (N=114)
Anaemia (Blood and lymphatic system disorders) | 6 | 3 | 12
Nausea (Gastrointestinal disorders) | 12 | 6 | 18
Diarrhoea (Gastrointestinal disorders) | 6 | 5 | 12
Vomiting (Gastrointestinal disorders) | 4 | 4 | 11
Abdominal pain (Gastrointestinal disorders) | 1 | 2 | 6
Constipation (Gastrointestinal disorders) | 1 | 1 | 6
Abdominal discomfort (Gastrointestinal disorders) | 2 | 3 | 2
Abdominal distension (Gastrointestinal disorders) | 0 | 0 | 6
Fatigue (General disorders) | 24 | 19 | 41
Irritability (General disorders) | 7 | 2 | 14
Pyrexia (General disorders) | 2 | 3 | 7
Upper respiratory tract infection (Infections and infestations) | 8 | 5 | 13
Bronchitis (Infections and infestations) | 1 | 4 | 11
Nasopharyngitis (Infections and infestations) | 3 | 0 | 10
Oral herpes (Infections and infestations) | 2 | 3 | 5
Herpes simplex (Infections and infestations) | 4 | 0 | 1
Decreased appetite (Metabolism and nutrition disorders) | 3 | 2 | 7
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 2 | 6
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 0 | 7
Headache (Nervous system disorders) | 9 | 5 | 16
Dizziness (Nervous system disorders) | 1 | 4 | 7
Insomnia (Psychiatric disorders) | 14 | 8 | 15
Depression (Psychiatric disorders) | 6 | 1 | 8
Anxiety (Psychiatric disorders) | 2 | 0 | 8
Cough (Respiratory, thoracic and mediastinal disorders) | 4 | 4 | 14
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 2 | 9
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 2 | 8
Respiratory tract congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 3 | 1
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 3 | 1
Rash (Skin and subcutaneous tissue disorders) | 3 | 4 | 7
Pruritus (Skin and subcutaneous tissue disorders) | 6 | 2 | 6
Dry skin (Skin and subcutaneous tissue disorders) | 2 | 0 | 6

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
After conclusion of the study and without prior written approval from Gilead, investigators in this study may communicate, orally present, or publish in scientific journals or other media only after the following conditions have been met:

* The results of the study in their entirety have been publicly disclosed by or with the consent of Gilead in an abstract, manuscript, or presentation form; or
* The study has been completed at all study sites for at least 2 years